CLINICAL TRIAL: NCT06154174
Title: Choline to Improve Malnutrition and Enhance Cognition
Acronym: CHIME-SAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Project Peanut Butter (Other); Kamuzu University of Health Sciences (Other); Balchem Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202308160
Record Dates: First submitted 2023-10-18; First posted 2023-12-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Severe Acute Malnutrition; Cognitive Impairment; Wasting; Kwashiorkor
MeSH Terms: conditions — Severe Acute Malnutrition; Cognitive Dysfunction; Cachexia; Kwashiorkor | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention and control RUTFs will be packaged in identical opaque sachets aside from colored stickers which will indicate randomization group. The intervention and control RUTFs will be identical in appearance, consistency, and smell. Efforts have been made to mask possible taste differences resulting from choline, including by the addition of a small amount (5mg) of choline to the control food. Participant masking cannot be guaranteed, however.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-RUTF (Ready-to-Use Therapeutic Food with added choline) (Experimental): A daily dose of 500mg choline will be added to RUTF. 2 sachets (daily dose) of RUTF will provide approximately 1000 Kcal, 14g of protein, 28g of fat, and 1 RDA of 14 micronutrients.
  Interventions: Dietary Supplement: C-RUTF (Ready-to-Use Therapeutic Food with added choline); Drug: Amoxicillin
- S-RUTF (Ready-to-Use Therapeutic Food without added choline) (Active Comparator): A daily dose of 5mg choline will be added to RUTF for masking. 2 sachets (daily dose) of RUTF will provide approximately 1000 Kcal, 14g of protein, 28g of fat, and 1 RDA or 14 micronutrients.
  Interventions: Dietary Supplement: S-RUTF (Ready-to-Use Therapeutic Food without added choline); Drug: Amoxicillin

INTERVENTIONS:
Dietary Supplement: C-RUTF (Ready-to-Use Therapeutic Food with added choline) — Choline added to peanut paste-based ready-to-use therapeutic food meeting Codex Alimentarius specifications
  Arms: C-RUTF (Ready-to-Use Therapeutic Food with added choline)
Dietary Supplement: S-RUTF (Ready-to-Use Therapeutic Food without added choline) — Standard peanut paste-based ready-to-use therapeutic food meeting Codex Alimentarius specifications
  Arms: S-RUTF (Ready-to-Use Therapeutic Food without added choline)
Drug: Amoxicillin — Oral amoxicillin tablets twice per day for 7 days dosed based on weight

SUMMARY:
The goal of this clinical trial is to test adding choline to ready-to-use therapeutic food (RUTF) in children with severe acute malnutrition (SAM) in Malawi. The main question it aims to answer is:

- Will the addition of a 500mg daily dose of choline to RUTF during treatment for SAM improve cognitive development among 6-59-month-old Malawian children compared with standard RUTF without added choline?

DETAILED DESCRIPTION:
Severe acute malnutrition (SAM) affects approximately 14 million children worldwide at any one time and has an annual incidence of 3-5x this number. SAM is defined by wasting (mid-upper arm circumference < 11.5 cm or weight-for-length z-score < -3) or presence of bilateral pedal pitting edema. SAM increases short-term risks for infection, hospitalization, and death, as well as longer-term risks for stunted linear growth and impaired cognitive development. This lattermost consequence is increasingly recognized, with studies showing that children who have suffered from SAM score 2-3 standard deviations below age-expected norms on cognitive development tests.

Ready-to-use therapeutic food (RUTF) revolutionized SAM treatment by allowing it to occur in the home setting. RUTF cures most children with SAM and ameliorates many of its worst consequences. RUTF was designed to be food-safe and promote anthropometric recovery. Since its inception, evidence has accumulated suggesting that the original fatty acid content of RUTF was not optimized for cognitive recovery from SAM. A 2021 trial, the Improved PUFA Trial (PMID: 34726694), demonstrated that reducing the omega-6 fatty acid content of RUTF and adding docosahexaenoic acid (DHA) improved cognitive development 6 months after SAM treatment in Malawian children. It is possible that further modifications to RUTF's composition might promote greater cognitive recovery.

Choline is essential for human health and development and is recognized as such by the Institute of Medicine, which designates daily recommended intakes. Choline deficiency has been shown to induce a host of cognitive developmental problems in animal models, is associated with neural tube defects in humans, and mutations of choline transporters in humans yield developmental degenerative conditions which, while rare, shed light on the essential nature of choline in brain development. Several small randomized, controlled trials have shown benefits of choline supplementation during early life on child cognitive development, both in healthy children and in those exposed to insults such as in fetal alcohol syndrome.

Choline plays important roles in brain structure and function and is found primarily in animal-source foods, which are deficient in the diets of children with SAM. Choline is an essential component of the neuronal membrane as well as a precursor for acetylcholine, a key neurotransmitter. In addition, choline plays a role in the trafficking and cell membrane integration of DHA, which rapidly accumulates in the human brain during childhood and ultimately composes 40-50% of brain polyunsaturated fatty acids. Decades of findings from epidemiological studies and laboratory science, including with animal models, support the essential role of DHA in the structure and function of the brain and retina. The Improved PUFA Trial leveraged these insights and showed that the developing brain is sensitive to fatty acid intake in the context of SAM; providing DHA in RUTF improved brain development. Hepatic export of DHA into plasma and its target tissues, including the brain, relies in part on synthesis of phosphatidylcholine (PC) by phosphatidylethanolamine N-methyltransferase (PEMT). DHA-enriched PC molecules (PC-DHA) are generated by PEMT and exported for delivery throughout the body. Indeed, PEMT-deficient mice have reduced DHA plasma concentrations and pups born to PEMT-deficient dams have limited DHA brain accumulation. The PEMT pathway relies on adequate supply of dietary methyl donors such as choline. Pairing (1) choline's ability to increase DHA trafficking to/integration within the brain with (2) the power of DHA in SAM, it is possible that adding choline to RUTF containing DHA might promote cognitive recovery and development among malnourished children.

This will be an individually randomized, investigator/outcomes assessors/caregiver-blinded, controlled clinical trial designed to determine whether the addition of a daily dose of 500mg of choline to ready-to-use therapeutic food (C-RUTF) will improve cognitive development among Malawian children 6-59 months of age with SAM compared with standard RUTF (S-RUTF). This trial will be conducted at 10 rural sites in southern Malawi. 1500 children will be randomized 1:1 to receive 2 sachets per day of either C-RUTF or S-RUTF. Children will receive their allocated RUTF and return to clinic fortnightly for repeat anthropometric measurements, illness questions, and to receive more RUTF until they achieve a clinical outcome or for a maximum of 12 weeks, at which point they will undergo Malawi Developmental Assessment Tool (MDAT) testing and blood spot collection. Participants will be asked to return to clinic 5-7 months later for MDAT testing, the global z-score from which will be the trial's primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 6-59 months of age
* mid-upper arm circumference < 11.5 cm and/or weight-for-length z-score < -3 and/or presence of bilateral pedal pitting edema
* willingness to comply with all study procedures and availability for the duration of the study, including no plan to move from the catchment area of a participating clinic

Exclusion Criteria:

* features of complicated SAM: inability to tolerate a 30g test dose of RUTF, breathing difficulties, mental status changes, sepsis, or physician/nursing clinical assessment that the child needs immediate hospitalization
* participation in a separate feeding program within the past month
* known allergy to study food ingredient (peanut, milk, fish)
* intention to move away from catchment area within 9 months
* developmental delay
* presence of a chronic severe medical condition (other than TB and HIV), such as congenital heart disease

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Malawi Developmental Assessment Tool global z-score | 6 months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better

SECONDARY OUTCOMES:
Malawi Developmental Assessment Tool gross motor sub-domain z-score | 6 months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor sub-domain z-score | 6 months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language sub-domain z-score | 6 months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social sub-domain z-score | 6 months after SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool global z-score | Within 1 month of SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool gross motor sub-domain z-score | Within 1 month of SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool fine motor sub-domain z-score | Within 1 month of SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool language sub-domain z-score | Within 1 month of SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Malawi Developmental Assessment Tool social sub-domain z-score | Within 1 month of SAM outcome
  Age-standardized score, -6 to +6, higher scores are better
Recovery | 2-12 weeks of therapeutic feeding
  Defined based on enrollment (anthropometric +/- edema) criteria
DHA status | 2-12 weeks of therapeutic feeding (until SAM outcome)
  Blood spot DHA % of total fatty acids in subset of participants
Time-to-recovery | 2-12 weeks of therapeutic feeding
  Weeks until recovery criteria met, with recovery defined based on enrollment criteria
Proportion of participants who die | 2-12 weeks of therapeutic feeding
  Defined by caregiver report
Proportion of participants who die | From enrollment to study end (6-month post-SAM-outcome MDAT visit)
  Defined by caregiver report
Proportion of participants remaining with SAM | After 12 weeks of therapeutic feeding
  Continue to meet SAM criteria after feeding
Proportion of participants with kwashiorkor resolution | 2-12 weeks of therapeutic feeding
  Resolution of nutritional edema
Time-to-kwashiorkor resolution | 2-12 weeks of therapeutic feeding
  Time to resolution of nutritional edema
Rate of weight gain | 2-12 weeks of therapeutic feeding (until SAM outcome)
  g/kg/day
Rate of length gain | 2-12 weeks of therapeutic feeding (until SAM outcome)
  mm/week
Proportion of participants with recurrence of SAM | From recovery until study end (6-month post-SAM-outcome MDAT visit)
  After recovery, again meeting criteria for SAM
Change in MDAT global z-score | From MDAT near time of SAM outcome to 6-month post-SAM-outcome MDAT visit
  Difference in MDAT global z-score between 6-month post-SAM outcome visit and MDAT, global z-score measured within 1 month of SAM outcome, more positive scores are better
Proportion of participations requiring hospitalization | Enrollment to 6-month post-SAM-outcome MDAT visit)
  Safety outcome
Diarrhea | 2-12 weeks of therapeutic feeding (until SAM outcome)
  Days, reported by caregiver, safety outcome

OTHER OUTCOMES:
MDAT global z-score by age | 6-month post-outcome MDAT visit
  Subgroups: enrollment <12 vs. >=12 months of age, -6 to +6, higher scores are better
MDAT global z-score by SAM outcome status | 6-month post-outcome MDAT visit
  Subgroups: Recovered vs. Other, -6 to +6, higher scores are better

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (10):
- Malawi (10):
  - Makhwira, Makhwira, Chikwawa
  - Mitondo, Mitondo, Chikwawa
  - Nkhate, Nkhate, Chikwawa
  - Chipolonga, Chipolonga, Machinga
  - Chikonde, Chikonde, Mulanje
  - Mbiza, Mbiza, Mulanje
  - Milonde, Milonde, Mulanje
  - Muloza, Muloza, Mulanje
  - Namasalima, Namasalima, Mulanje
  - Naphimba, Naphimba, Mulanje

IPD SHARING:
Plan to Share IPD: Yes
All collected, de-identified individual patient data
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within 12 months of primary publication